CLINICAL TRIAL: NCT00589108
Title: A Prospective, Randomized, Controlled Study Comparing A Mobile-Bearing Total Knee System With A Fixed-Bearing Total Knee System In Cemented Total Knee Arthroplasty
Brief Title: Comparison of A Mobile-Bearing Total Knee System With A Fixed-Bearing Total Knee System In Cemented Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert T. Trousdale, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 271-01
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2012-12

CONDITIONS: Degenerative Joint Disease
Keywords: knee arthroplasty
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobile-Bearing Knee (Active Comparator): Sigma Knee System (mobile-bearing knee with the P.S. polyethylene insert)
  Interventions: Device: Sigma Knee System
- Modular-Metal-Backed Knee (Active Comparator): Sigma Pressfit Condylar Posterior Cruciate Substituting System with a metal back tibial tray (fixed-bearing knee with the metal backed tray)
  Interventions: Device: Sigma Pressfit Condylar Posterior Cruciate Substituting System with a metal back tibial tray
- All-Polyethylene Knee (Active Comparator): Sigma Pressfit Condylar Posterior Cruciate Substituting System all polyethylene tray
  Interventions: Device: Sigma Pressfit Condylar Posterior Cruciate Substituting System all polyethylene tray

INTERVENTIONS:
Device: Sigma Knee System — Sigma Knee System (mobile-bearing knee with the P.S. polyethylene insert)
  Other Names: Sigma Rotating Platform Knee System
  Arms: Mobile-Bearing Knee
Device: Sigma Pressfit Condylar Posterior Cruciate Substituting System with a metal back tibial tray — Sigma Pressfit Condylar Posterior Cruciate Substituting System with a metal back tibial tray (fixed-bearing knee with the metal backed tray)
  Other Names: Press-Fit Condylar Total Knee Arthroplasty
  Arms: Modular-Metal-Backed Knee
Device: Sigma Pressfit Condylar Posterior Cruciate Substituting System all polyethylene tray — Sigma Pressfit Condylar Posterior Cruciate Substituting System (fixed bearing with an all polyethylene tray)
  Arms: All-Polyethylene Knee

SUMMARY:
Pain, weakness, instability, and progressive dysfunction are the hallmarks of arthritis of the knee. Total knee replacement may frequently be the only therapeutic intervention to provide adequate improvement in pain and function. Both fixed bearing and mobile bearing knees have a long track record of clinical success. Mobile bearing designs have theoretical advantages of decreased contact stresses on the tibial tray, decreased polyethylene wear, and improved range of motion relative to fixed bearing designs. These theoretical advantages may become especially important in the young patient who requires a knee arthroplasty. This study will attempt to see if there is a clinical difference in outcome between mobile bearing and fixed bearing knee arthroplasties in patients who require total knee replacement.

DETAILED DESCRIPTION:
This prospective, randomized, single-blinded clinical trial compared a mobile-bearing total knee system with two types of fixed-bearing total knee systems in patients undergoing cemented total knee arthroplasty. The devices to be used are FDA approved: the Sigma Knee System (mobile-bearing), the Sigma, Pressfit Condylar posterior cruciate substituting (fixed-bearing) system with a metal backed tibial tray, and the Sigma press-fit condylar posterior cruciate substituting system (fixed bearing) with an all polyethylene tibial tray.

The surgical procedures were performed by 4 experienced orthopedic surgeons with a subspecialty interest in total knee arthroplasty. A midline skin incision and medial parapatellar arthrotomy were used to expose the knee. The distal femoral resection was performed with an intramedullary alignment guide, and the proximal tibial resection was performed with an extramedullary alignment guide. Knees with fixed deformities had a surgical release of the contracted tissues on the medial or lateral side, as appropriate, to obtain symmetric balance of the total knee replacement in both flexion and extension. The flexion and extension gaps and the medial and lateral soft-tissue structures were balanced in accordance with standard techniques.

Patients began progressive weight-bearing on the first postoperative day, and active knee range of motion was initiated with 24 hours after surgery. Patients were typically discharged on the fourth or fifth postoperative day after obtaining the ability to walk with a walker, to ascend several stairs, and to flex the knee 290 degrees. Patients were asked to return for examination and radiographs at 3 months, 1 year, 2 years, and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary knee surgery for degenerative joint disease (DJD).

Exclusion Criteria:

* Severe deformity greater than or equal to 20 degrees varus, valgus malalignment
* Osteomyelitis, septicemia, or other active infections that may spread to other areas of the body
* The presence of infections, highly communicable diseases, e.g., AIDS, active tuberculosis, venereal disease, hepatitis
* Significant neurological or musculoskeletal disorders or disease that may adversely affect normal gait or weight bearing
* Metastatic disease
* Any congenital, developmental, or other bone disease or previous knee surgery that may, in the surgeon's judgement, interfere with total knee prosthesis survival or success, e.g., Paget's disease, Charcot's disease secondary to diabetes, severe osteoporosis, previous high tibial osteotomy, etc.
* Presence of previous prosthetic knee replacement device (any type)
* Arthrodesis of the affected knee
* Patients not requiring patella resurfacing.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2001-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Trousdale, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Kalisvaart MM, Pagnano MW, Trousdale RT, Stuart MJ, Hanssen AD. Randomized clinical trial of rotating-platform and fixed-bearing total knee arthroplasty: no clinically detectable differences at five years. J Bone Joint Surg Am. 2012 Mar 21;94(6):481-9. doi: 10.2106/JBJS.K.00315. PMID 22437996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study began on March 1, 2001, and continued through March 1, 2003.
Pre-assignment Details: 397 subjects were assessed for eligibility and 157 were excluded prior to randomization because they either declined to participate (n=53), or did not meet inclusion criteria (n=104).
Period: Overall Study
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Started | 80 | 80 | 80
Completed | 76 | 76 | 75
Not Completed | 4 | 4 | 5
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Death | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee | Total
Number analyzed (Participants) | 80 | 80 | 80 | 240
Age Continuous [Median (Full Range); unit: years] | 69.0 [41 to 81] | 68.5 [41 to 81] | 69.0 [41 to 81] | 68.5 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 55 | 167
  Male | 24 | 24 | 25 | 73
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 80 | 240

OUTCOME MEASURES:

1. Primary Outcome: Maximum Knee Flexion
Description: The range of knee motion was measured clinically with use of a goniometer. Measurements were performed by physician assistants in the Department of Orthopedic Surgery who were blinded to the type of implant used. The subject was positioned supine on the examination table, and maximum active flexion was measured.
Time Frame: 2 years post-surgery, 5 years post-surgery
Measure: Mean (Full Range); unit: degrees
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Number analyzed (Participants) | 76 | 76 | 75
degrees
  2 years post-surgery | 110 [90 to 130] | 111 [90 to 130] | 111 [90 to 140]
  5 years post-surgery | 109.0 (15.27) [40 to 140] | 109 (14.28) [60 to 140] | 110.0 (13.75) [80 to 140]
Statistical Analysis 1: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference between the mean maximum flexion between the three groups at 2 years post-surgery; Test type: Superiority or Other; p = 0.64, ANOVA
Statistical Analysis 2: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference between the mean maximum flexion between the three groups at 5 years post-surgery; Test type: Superiority or Other; p = 0.80, ANOVA

2. Secondary Outcome: Knee Society Function Score
Description: The Knee Society Function Score considers only walking distance and stair climbing, with deductions for walking aids. The maximum function score, which is 100, is obtained by a patient who can walk an unlimited distance and go up and down stairs normally. The minimum function score is 0.
Time Frame: 5 years post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Number analyzed (Participants) | 76 | 76 | 75
units on a scale | 69.2 (23.44) | 77.4 (23.44) | 69.7 (26.09)
Statistical Analysis 1: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference for the Knee Society Function Score between the three groups at 5 years post-surgery; Test type: Superiority or Other; p = 0.06, ANOVA

3. Secondary Outcome: Knee Society Pain Score
Description: The Knee Society Pain Score includes walking and climbing stairs. The maximum score per knee is 50 indicating no pain, and 0 indicates severe pain. Therefore the total score (for both knees) could range from 0 to 100.
Time Frame: 5 years post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Number analyzed (Participants) | 76 | 76 | 75
units on a scale | 87.8 (12.17) | 88.7 (9.93) | 88.3 (11.58)
Statistical Analysis 1: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference for the Knee Society Pain Score between the three groups at 5 years post-surgery; Test type: Superiority or Other; p = 0.87, ANOVA

4. Secondary Outcome: Knee Society Stair Climbing Score
Description: The stair-climbing portion of the Knee Society clinical rating system assigns a maximum score of 50 points for patients able to ascend and descend stairs in a normal fashion, 40 points for patients needing a rail to descend, 30 points for patients using a rail in both directions, 15 points for patients able to ascend but not descend at all, and 0 points for patients unable ascend or descend. Because stair ascent and descent put substantial demands on the patellofemoral joint, we used that portion of the Knee Society clinical rating system as a proxy for patellofemoral function in this study.
Time Frame: two years post-surgery, five years post-surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Number analyzed (Participants) | 76 | 76 | 75
units on a scale
  Two years post-surgery | 39 [0 to 50] | 40 [0 to 50] | 39 [0 to 50]
  Five years post-surgery | 36 [0 to 50] | 40 [0 to 50] | 37 [0 to 50]
Statistical Analysis 1: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference between the Knee Society Stair Climbing Score between the three groups at 2 years post-surgery; Test type: Superiority or Other; p = 0.44, ANOVA
Statistical Analysis 2: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference between the Knee Society Stair Climbing Score between the three groups at 5 years post-surgery; Test type: Superiority or Other; p = 0.08, ANOVA

5. Secondary Outcome: Percentage of Knees Surviving at 5 Years
Description: Kaplan-Meier analysis of five-year implant survival rate
Time Frame: 5 years post-surgery
Measure: Number; unit: percentage of knees
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Number analyzed (Participants) | 76 | 76 | 75
percentage of knees
  With revision for any reason as end point | 98.7 | 97.4 | 98.7
  With revision for aseptic loosening as end point | 100 | 97.4 | 98.7
Statistical Analysis 1: Comparison: Mobile-Bearing Knee vs Modular-Metal-Backed Knee vs All-Polyethylene Knee; P-value for the difference between the percentage of knees surviving between the three groups at 5 years post-surgery; Test type: Superiority or Other; p = 0.92, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 5 years that the subjects were on the study.
Arm/Group | Mobile-Bearing Knee | Modular-Metal-Backed Knee | All-Polyethylene Knee
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 5/76 | 4/76 | 2/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobile-Bearing Knee (N=76) | Modular-Metal-Backed Knee (N=76) | All-Polyethylene Knee (N=75)
Aseptic loosening (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Patellar crepitus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Knee stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No